CLINICAL TRIAL: NCT03694782
Title: Community Gardens Participation in Promoting Sustainable Lifestyles in Urban Settings: the JArDinS Study
Status: Completed | Type: Observational
Sponsor: Institut National de Recherche pour l'Agriculture, l'Alimentation et l'Environnement (Other)
Responsible Party: Principal Investigator, Marion Tharrey, Principal investigator, Institut National de Recherche pour l'Agriculture, l'Alimentation et l'Environnement
Other Study IDs: JArDinS
Record Dates: First submitted 2018-09-25; First posted 2018-10-03 (Actual); Last update posted 2020-02-11 (Actual); Status verified 2020-02

CONDITIONS: Sustainable Lifestyles
Keywords: diet; food prices; environment; physical activity; nature; well being; natural experiment; loneliness; accelerometry
MeSH Terms: conditions — Motor Activity | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Experimental group: Gardeners starting gardening in a community garden in Montpellier (France)
  Interventions: Behavioral: Food diary supply; Behavioral: Actigraph; Behavioral: Questionnaire
- Control Group: Volunteers living in the same neighborhoods but with no experience in community gardening.
  Interventions: Behavioral: Food diary supply; Behavioral: Actigraph; Behavioral: Questionnaire

INTERVENTIONS:
Behavioral: Food diary supply — Each participant was issued with a food supply diary to record details of their household food supply and related trips over 1-mo period. Household food supply included food purchases, food gift/donation, and potential crops from the garden. Away-from-home food consumption was not recorded. For each food purchase, participants provided details of date, place of purchase, foods purchased (name, quantity and expense incurred), and trip made (origin/where the trip started, destination/where the trip ended, and mode of transportation). When till receipts were available in grocery stores or supermarkets, participants were asked to collect them in an envelope placed at the end of the food supply diary. To facilitate data entry, all family members were encouraged to help filling out the diary.
Behavioral: Actigraph — Participants were instructed to wear a triaxial accelerometer (wGT3X-BT or wActiSleep-BT, Actigraph, Pensacola, FL, USA) fitted with an elastic strap on right side of the hip for 9 consecutive days, except for bathing and performing activities in the water. The Actigraph was accompanied by an activity logbook in which participants were required to daily record time when awake and sleeping, and, if any, time and duration of workout or device removal
Behavioral: Questionnaire — Participants received by email a link to complete an online questionnaire about mental and social health, sensibility to food waste, and connection with nature

SUMMARY:
The JArDinS study is a quasi-experimental research that aimed at assessing the impact of community garden participation (a natural experiment) in the adoption of more sustainable lifestyles.

DETAILED DESCRIPTION:
The JArDinS study is part of the SURFOOD-Foodscapes project evaluating the relationships between urban foodscape and food styles in Montpellier Metropole (France).

JArDinS consists of a pretest-posttest quasi-experimental research and includes an experimental group of new gardeners starting gardening in a community garden in Montpellier and a control group comprising participants from a survey on food behaviors undertaken as part of SURFOOD-Foodscapes project. Participants will be surveyed at enrollment and 12 months later.

ELIGIBILITY:
Inclusion Criteria:

* starting gardening in a community garden (for experimental group)
* no experience in community gardening (for control group)
* willingness to be involved in the study through one year
* age above 18 years
* ability to read in French and live in the city of Montpellier.

Exclusion Criteria:

* past experience of at least one household member in community gardening
* never doing grocery shopping for home

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: residents of Montpellier (France)
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2020-02-10 (Actual); Study Completion 2020-02-10 (Actual)

PRIMARY OUTCOMES:
Change in healthiness of household food supply | at baseline and exactly 12 month later
  The nutritional quality of household food supply was estimated using two indicators of nutritional quality : the mean adequacy ratio (MAR) and the mean excess ratio (MER)
Change in physical activity energy | at baseline and exactly 12 month later
  Physical activity energy expenditure were estimated directly from raw triaxial accelerometry data using a model which combines an automatic activity-recognition algorithm with an activity-specific count-based model
Change in mental well-being | at baseline and exactly 12 month later
  Assessed by the Warwick-Edinburgh Mental Wellbeing Scale. WEMWBS is a 14-item scale rated on a 5-point Likert-type, in which all items are worded positively and address aspects of positive mental health. Total score range from 14-70, with higher scores indicating a higher level of mental well-being.
Change in social isolation | at baseline and exactly 12 month later
  Assessed by the UCLA Loneliness Scale. UCLA-3 is a 20-item scale (11 positive and 9 negative) rated on a 4-point Likert-type. Total score range from 20-70, with higher scores greater feelings of loneliness.
Change in environmental impact of household's food supply | at baseline and exactly 12 month later
  Greenhouse gas emissions (in g CO2eq), atmospheric acidification (g SO2eq) and marine eutrophication (in g Neq) related to household's food supply were computed using estimates from the French 'SUStable' table.
Change in environmental impact of household's food trip (in g CO2eq) | at baseline and exactly 12 month later
  For each food trip, the distance traveled specifically for food purchase will be multiplied by energy source consumption of the transportation used, and by the corresponding GHGE factor of source consumption. GHGE related to food trip will be calculated as the sum of all food trips during the period of data collection.
Change in sensibility to food waste | at baseline and exactly 12 month later
  Assessed by the Sensibility to food waste scale, a 8-item scale rated on a 7-point Likert-type, that measure in which extent participants attach importance to waste and are emotionally affected by it. Total score range from 7-56, a higher total scores denote greater sensibility to food waste.
Change in connection with nature | at baseline and exactly 12 month later
  Affective, cognitive, and experiential aspects of individuals' connection to nature was assessed by the Nature Relatedness Scale (NRS). NRS is a 21-item scale rated on a 5-point Likert-type. Total score range from 5-105, a higher total scores denote greater nature connectedness.
Change in household food supply expenditure | at baseline and exactly 12 month later
  Monthly household food expenditure and the contribution of each food group and subgroup to total food expenditure were estimated using food expenses data collected in the food supply diary.

SECONDARY OUTCOMES:
Age (in year) of each member of the household | at baseline
  Participants were asked to report the age of each member each adult of the household.
Gardening experience prior to the project | at baseline
  Participants were asked about their experiences and perceived competence in gardening.
Gender of each member of the household | at baseline
  Participants were asked to report the gender of each adult of the household
Household income | at baseline
  Participants indicated their net income bracket of the household (by month).
Education level of each adult of the household | at baseline
  Participants were asked to report the higest education level achieved by each adult of the household.

CONTACTS AND LOCATIONS:
Locations (1):
- INRA, Montpellier, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tharrey M, Sachs A, Perignon M, Simon C, Mejean C, Litt J, Darmon N. Improving lifestyles sustainability through community gardening: results and lessons learnt from the JArDinS quasi-experimental study. BMC Public Health. 2020 Nov 26;20(1):1798. doi: 10.1186/s12889-020-09836-6. PMID 33243204
- [Derived] Tharrey M, Perignon M, Scheromm P, Mejean C, Darmon N. Does participating in community gardens promote sustainable lifestyles in urban settings? Design and protocol of the JArDinS study. BMC Public Health. 2019 May 17;19(1):589. doi: 10.1186/s12889-019-6815-0. PMID 31101095